CLINICAL TRIAL: NCT05933707
Title: Effect of Small Extracellular Vesicles From Adipose Tissue on Insulin Action
Brief Title: Small Extracellular Vesicles and Insulin Action
Acronym: SEV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 202005117
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Obesity; Insulin Resistance; Metabolically Healthy Obesity; Obesity, Metabolically Benign
Keywords: Obesity; Weight Loss; Exosomes; Extracellular vesicles
MeSH Terms: conditions — Obesity; Insulin Resistance; Obesity, Metabolically Benign; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Metabolically healthy lean - Baseline testing only (No Intervention): Metabolically healthy lean - Lean individuals that have good glucose (sugar) control (defined as normal fasting glucose, glucose tolerance and hemoglobin A1c), normal insulin sensitivity (defined as Homeostatic Model Assessment of Insulin Resistance [HOMA-IR] <2.5) and normal intrahepatic triglyceride (fat) levels.
  Dietary intervention - None.
- People with Metabolically Healthy Obesity - Baseline testing only (No Intervention): People with Metabolically Healthy Obesity - Persons with obesity that have good glucose (sugar) control, normal insulin sensitivity and normal intrahepatic triglyceride (fat) levels.
  Dietary intervention - None.
- People with Metabolically Unhealthy Obesity - Low Calorie Diet (Experimental): People with Metabolically Unhealthy Obesity - Persons with obesity with plasma glucose and intrahepatic triglyceride (fat) levels higher than recommended in combination with insulin resistance (defined as HOMA-IR ≥2.5).
  Dietary intervention - Low calorie diet.
  Interventions: Behavioral: People with Metabolically Unhealthy Obesity - Low Calorie Diet

INTERVENTIONS:
Behavioral: People with Metabolically Unhealthy Obesity - Low Calorie Diet — Consumption of a low-calorie diet with caloric intake reduced by ~25% to achieve ~10% weight loss in about 4 to 5 months.
  Other Names: Dietary weight loss
  Arms: People with Metabolically Unhealthy Obesity - Low Calorie Diet

SUMMARY:
The goals of this research study are to: 1) understand why some people with obesity are protected from developing conditions such as type 2 diabetes and cardiovascular disease while others are more likely to develop obesity-related conditions; 2) assess the effect of small extracellular vesicles (sEVs also called exosomes), obtained from human participants, on metabolic function in cultured cells and in mice.

DETAILED DESCRIPTION:
Insulin resistance is commonly associated with obesity and is a major contributor to the development of obesity-related metabolic diseases, including nonalcoholic fatty liver disease, the metabolic syndrome, and type 2 diabetes (T2D). Most persons with obesity are "metabolically unhealthy" (MUO), often defined by having insulin resistance and the metabolic syndrome. However, a subset of people with obesity are metabolically healthy (MHO) and protected from the adverse metabolic effects of excess adiposity. The mechanisms that determine the differences in metabolic health between people with MUO and MHO are not unclear. This project will examine the effects of plasma and adipose tissue small extracellular vesicles (sEVs) on multi-organ insulin action. The investigators will isolate sEVs from subcutaneous abdominal adipose tissue biopsies and blood samples obtained from human participants with MHO, MUO or who are metabolically healthy and lean (MHL) and examine the effects of these sEVs on insulin resistance in muscle, liver and fat cells in culture and on multi-organ insulin sensitivity in lean and obese mice. The investigators will also identify differences in the potential bioactive molecules, namely miRNA and bioactive lipids, that are carried by sEVs. The results from this study will help determine whether plasma or adipose tissue sEVs in people who are MHL, MHO, or MUO are involved in regulating liver, muscle and adipose tissue insulin sensitivity. These results could identify novel pathways that regulate metabolic health in people and provide the foundation for exploring the potential of sEVs as a therapeutic target to prevent and treat the metabolic complications of obesity.

ELIGIBILITY:
Inclusion Criteria:

* Metabolically healthy lean subjects must have a BMI ≥18.5 and ≤24.9 kg/m²; Subjects with obesity must have a BMI ≥30.0 and ≤50.0 kg/m²
* Metabolically healthy lean and people with metabolically healthy obesity must have intrahepatic triglyceride (IHTG) content ≤5%; fasting plasma glucose concentration <100 mg/dl, 2-hr oral glucose tolerance plasma glucose concentration <140 mg/dl, hemoglobin A 1C (HbA1c) ≤5.6% and HOMA-IR <2.5.
* People with metabolically unhealthy obesity must have intrahepatic triglyceride (IHTG) content ≥5.6%; HOMA-IR ≥2.5, and HbA1c 5.7%-6.4%, or fasting plasma glucose concentration ≥100 mg/dl, or 2-hr oral glucose tolerance test (OGTT) plasma glucose concentration ≥140 mg/dl.

Exclusion Criteria:

* History of diabetes, liver disease other than NAFLD or other serious diseases,
* Consume excessive amounts of alcohol (>21 units/week for men and >14 units/week for women),
* Take medications that could affect the study outcome measures, engage in regular exercise (>120 min/week),
* Are pregnant or lactating

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-06-08 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Effect of exosomes on insulin sensitivity in cultured cells | Baseline only (cross-sectional comparison of metabolically healthy lean, and of people with metabolically healthy or metabolically unhealthy obesity).
  Exosomes obtained from the plasma and adipose tissue of metabolically healthy lean participants, and participants with metabolically healthy or metabolically unhealthy obesity will be tested in cultured cells and mice to determine their effect on insulin sensitivity.
Change in the effect of exosomes on insulin sensitivity | Before and after ~10% weight loss (~4-5 months) in people with metabolically abnormal obesity
  Exosomes obtained from the plasma and adipose tissue of participants with metabolically unhealthy obesity before and after 10% weight loss will be tested in cultured cells and mice to determine their effect on insulin sensitivity.

SECONDARY OUTCOMES:
Differences in the content of microRNAs within exosomes obtained from plasma and adipose tissue | Baseline only (cross-sectional comparison of metabolically healthy lean, and of people with metabolically healthy or metabolically unhealthy obesity).
  Exosomes obtained from the plasma and adipose tissue of metabolically healthy lean participants, and participants with metabolically healthy or metabolically unhealthy obesity will be analyzed to determine their microRNA composition.
Differences in the content of lipids within exosomes obtained from plasma and adipose tissue | Baseline only (cross-sectional comparison of metabolically healthy lean, and of people with metabolically healthy or metabolically unhealthy obesity).
  Exosomes obtained from the plasma and adipose tissue of metabolically healthy lean participants, and participants with metabolically healthy or metabolically unhealthy obesity will be analyzed to determine their lipid composition.
Changes in the content of microRNAs within exosomes obtained from plasma and adipose tissue | Before and after ~10% weight loss (~4-5 months) in people with metabolically abnormal obesity
  Exosomes obtained from the plasma and adipose tissue of metabolically unhealthy obesity before and after weight loss will be analyzed to determine changes in their microRNA content after weight loss.
Changes in the content of lipids within exosomes obtained from plasma and adipose tissue | Before and after ~10% weight loss (~4-5 months) in people with metabolically abnormal obesity
  Exosomes obtained from the plasma and adipose tissue of metabolically unhealthy obesity before and after weight loss will be analyzed to determine changes in their lipid content after weight loss.
Insulin sensitivity | Baseline only (cross-sectional comparison of metabolically healthy lean, and people with metabolically healthy or metabolically unhealthy obesity).
  Whole-body insulin sensitivity will be assessed by using the hyperinsulinemic-euglycemic clamp procedure
Change in insulin sensitivity | Before and after ~10% weight loss (~4-5 months) in people with metabolically abnormal obesity
  Whole-body insulin sensitivity will be assessed by using the hyperinsulinemic-euglycemic clamp procedure
Fat mass and fat free mass | Baseline only (cross-sectional comparison of metabolically healthy lean, and people with metabolically healthy or metabolically unhealthy obesity).
  Fat mass and fat free mass will be assessed using dual-energy x-ray absorptiometry (DXA)
Change in fat mass and fat free mass | Before and after 10% weight loss (~4-5 months) in people with metabolically abnormal obesity
  Fat mass and fat free mass will be assessed using dual-energy x-ray absorptiometry (DXA)
Abdominal adipose tissue volumes | Baseline only (cross-sectional comparison of metabolically healthy lean, and people with metabolically healthy or metabolically unhealthy obesity).
  Abdominal subcutaneous and intra-abdominal adipose tissue volumes will be assessed by magnetic resonance imagining (MRI)
Change in abdominal adipose tissue volumes | Before and after ~10% weight loss (~4-5 months) in people with metabolically abnormal obesity
  Abdominal subcutaneous and intra-abdominal adipose tissue volumes will be assessed by magnetic resonance imagining (MRI)
Intra-hepatic triglyceride content | Baseline only (cross-sectional comparison of metabolically healthy lean, and people with metabolically healthy or metabolically unhealthy obesity).
  Intra-hepatic triglyceride content will be assessed by magnetic resonance techniques
Change in intra-hepatic triglyceride content | Before and after ~10% weight loss (~4-5 months) in people with metabolically abnormal obesity
  Intra-hepatic triglyceride content will be assessed by magnetic resonance techniques

CONTACTS AND LOCATIONS:
Overall Officials: Dmitri Samovski, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Currently there is no plan to share individual participant data.